CLINICAL TRIAL: NCT07144579
Title: Evaluation of the Effect of Music Listening on Pain, Anxiety, and Behavior in Children With Dental Anxiety During the Restoration of Permanent First Molars
Brief Title: Effect of Music on Pain, Anxiety, and Behavior in Anxious Children During Molar Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Elif UĞURBEKLER HÜNDÜ, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MersinU-DHF-EUH-01
Record Dates: First submitted 2025-08-14; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healhty
Keywords: cortisol; dental anxiety; children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): no audio distraction
- Mozart Music Group (Active Comparator): "Mozart - Sonata for Two Pianos in D, K. 448" music was played
  Interventions: Behavioral: Mozart music group
- Preferred music group (Active Comparator): The patient's requested music was played
  Interventions: Behavioral: preferred music group

INTERVENTIONS:
Behavioral: Mozart music group — The experimental group was played Mozart - Sonata for Two Pianos in D, K. 448 on the clinic computer.
  Arms: Mozart Music Group
Behavioral: preferred music group — The experimental group was made to listen to their preferred music in the clinic.
  Arms: Preferred music group

SUMMARY:
Managing the child's behavior and anxiety is critical for the treatment in pediatric dentistry to be successful. Behavior management techniques aim to reduce the need for excessive and potentially unsafe medication use. Audio distraction is a non-intrusive distraction technique in which patients listen to music or a story during a stressful procedure. The success of the vocal distraction technique has been validated in medical settings, but insufficient literature exists to measure the potency of this technique for the pediatric population. The aim of this study is to reveal the effects of listening to music during dental treatment on the anxiety of 45 patients aged 7-10 years with dentist anxiety who applied to Mersin University Faculty of Dentistry Pediatric Dentistry clinic in 2024. The compliance of children who apply for routine examination and treatment by the researcher will be evaluated according to the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS), and if they score between 32-38, they will be invited to the study. Patients who agree to participate in the study will be divided into 3 groups.In the control group consisting of 15 pediatric patients, routine treatment will be performed without any distraction. In the 2nd group (intervention group consisting of 15 people), the patient will receive routine treatment accompanied by music by opening Mozart's Sonata for Two Pianos in D Major, K.448 on the computer in the clinic. In the 3rd group (intervention group consisting of 15 participants), patients will be asked what music they want to listen to and will be played music accordingly. Later, in order to evaluate the effect of the music listened to during dental treatment on anxiety, measurements will be taken at the routine appointment to show the anxiety state before, after and during the treatment. These measurements were determined as a result of literature review as the Children's Fear Research Program Dental Subscale (CFSS-DS), blood pressure, pulse, body temperature, oxygen saturation and salivary cortisol levels. Cortisol levels will be measured using the Cortisol Salivary Enzyme Linked Immunosorbent Assay (ELISA) Test Kit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who applied to the Department of Pediatric Dentistry, Faculty of Dentistry, Mersin University, between 01.08.2024 and 01.08.2025
* Patients with moderate anxiety, scoring 32-38 points on the dental subscale of the Children's Fear Survey Schedule - Dental Subscale (CFSS-DS)
* Voluntary participation of both the child and the parent in the study
* Patients with no previous dental experience
* Absence of any urgent dental condition requiring immediate intervention (e.g., pain, abscess, fistula)
* Systemically healthy patients
* No previous dental treatment experience
* Signed informed consent form by the parent/guardian
* Children aged between 7 and 10 years
* Patients with dentinal caries in the mandibular permanent first molar
* Patients whose treatment duration is expected to be approximately 30-45 minutes

Exclusion Criteria:

* Child and/or parent unwilling to participate in the study
* Failure to sign the informed consent form/written consent form
* Presence of any systemic disease
* Patients with low or high anxiety levels, scoring below 32 or above 38 on the dental subscale of the Children's Fear Survey Schedule - Dental Subscale (CFSS-DS)
* Patients with previous dental experience
* Children younger than 7 years or older than 10 years
* Caries in the mandibular permanent first molar requiring pulp therapy
* Presence of abscess or inflammation originating from the mandibular permanent first molar
* Absence of caries in the mandibular permanent first molar
* Teeth in which a dental dam cannot be applied

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
pre-treatment and post-treatment cortisol level | Values were measured on the day of treatment.
  The patient's pre-treatment and post-treatment cortisol levels were measured and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin Universty, Mersin, yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No